CLINICAL TRIAL: NCT02356731
Title: The Diagnosis and Management of Patients With Epilepsy: Nationwide, Multicenter Study of Recordings for the Diagnosis and Management of Patients With Epilepsy and Treatment With Levetiracetam in Daily Clinical Practice in Greece
Brief Title: LevetIracetam in Patients Being Treated for Epilepsy
Acronym: LIBERTY
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-LVT-EL-54
Record Dates: First submitted 2015-01-23; First posted 2015-02-05 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Epilepsy
Keywords: seizures,; quality of life
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Epilepsy is one of the most common neurological diseases.Approximately 53 million people suffering from chronic recurrent epilepsy in 1990 and that number increased about 58 million in 2005.

The annual incidence of epilepsy varies considerably in different epidemiological studies, ranging from 11 cases per 100,000 general population to 230 cases per 100,000 people.

To date there has been discovered the ideal Antiepileptic Drugs. The drug, ie, that are safe and effective, it has good daily administration frequency, easily administered from all roads, which has high bioavailability, which is not highly bound to proteins, and not holding inductive or inhibitory effect.

DETAILED DESCRIPTION:
There are broad-spectrum anticonvulsant, which means that a drug can be very effective for a patient, but may or may not regulate and increase the frequency of another crisis. Thus there remains now only to choose one among a number of drugs, the most appropriate.This study intends to register within 12 months clinical practice in Greek reality as regards the elements of diagnosis and management of patients with epilepsy and those who already are, or are part of treatment with levetiracetam.

The aims of this clinical study is to record data on

* the diagnosis
* The management of epilepsy in daily clinical practice in a sample of Greek population
* The monitoring of patients entering or already undergoing treatment with levetiracetam.
* The assessment of quality of life between visits of the study by using quality of life QOLIE-31 questionnaire
* The economic evaluation of the change in treatment from original to generic levetiracetam This is a data recording study and evaluation of treatment with levetiracetam. The study will take place in 15 antiepileptic centers throughout Greece. Researchers will have to successively record all incidents of patients (30 per center) with epilepsy, which are new diagnoses or already diagnosed and are treated with levetiracetam.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Males and Females
* Age> 6 years
* Patients diagnosed with epilepsy or
* Patients who are diagnosed and treated with antiepileptic treatment levetiracetam
* Patients who consent to their participation in the study
* Patients will comply with the requirements and procedures of the study

Exclusion Criteria:

* Patients who did not consent to their participation in the study
* Patients who will not comply to the needs and the design process

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit outpatients who are new epilepsy diagnoses or diagnosed prior to enrollment in the study and treated with levetiracetam for the management of their disease. All patients will be included from 15 research centers nationwide. Each center will include ≥30 patients to be monitored (1: 1 newly diagnosed / older diagnoses).
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in seizures' status (Change of number of seizures from baseline) | 12 months
  Change of number of seizures from baseline

SECONDARY OUTCOMES:
Change in adverse events | 12 months
  Change of number of adverse events from baseline
Change in treatment cost | 12 months
  Change in treatment cost from baseline
Change in Quality of Life | 12 months
  Change in QoLie score from baseline

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Gennimatas General State Hospital, Athens, Attica
  - Papageorgiou Hospital, Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hauser WA. Recent developments in the epidemiology of epilepsy. Acta Neurol Scand Suppl. 1995;162:17-21. doi: 10.1111/j.1600-0404.1995.tb00493.x. PMID 7495183
- [Background] Sander JW, Shorvon SD. Epidemiology of the epilepsies. J Neurol Neurosurg Psychiatry. 1996 Nov;61(5):433-43. doi: 10.1136/jnnp.61.5.433. No abstract available. PMID 8965090
- [Result] Piperidou H, Terzoudi A, Vorvolakos T, Davis E, Heliopoulos I, Vadikolias K, Giassakis G, Aggelopoulos P, Georgios G, Karlovasitou A. The Greek version of the Quality of Life in Epilepsy Inventory (QOLIE-31). Qual Life Res. 2006 Jun;15(5):833-9. doi: 10.1007/s11136-005-5149-9. PMID 16721643
- [Result] 3. Hauser WA. Incidence and prevalence. In: ENGEL J Jr., PEDLEY A eds. Epilepsy: a comprehensive textbook. Philadelphia: Lippincot-Raven Publishers, 1997; 47-57
- [Result] ILAE Commission Report. The epidemiology of the epilepsies: future directions. International League Against Epilepsy. Epilepsia. 1997 May;38(5):614-8. No abstract available. PMID 9184609
- [Result] Hart YM, Sander JW, Johnson AL, Shorvon SD. National General Practice Study of Epilepsy: recurrence after a first seizure. Lancet. 1990 Nov 24;336(8726):1271-4. doi: 10.1016/0140-6736(90)92960-p. PMID 1978114
- [Result] 8. ENGEL J Jr. The epilepsies. In: Wyngaarden JB, Smith LH, Claude Bennet J (eds) Cecil Textbook of Medicine. Saunders, Philadelphia, 1992:2202-2213
- [Result] Triantafyllou NI, Zalonis I, Kokotis P, Anthracopoulos M, Siafacas A, Malliara S, Hamburger HL, Papageorgiou C. Cognition in epilepsy: a multichannel event related potential (P300) study. Acta Neurol Scand. 1992 Nov;86(5):462-5. doi: 10.1111/j.1600-0404.1992.tb05124.x. PMID 1481627
- [Result] Trimble MR. Anticonvulsant drugs and cognitive function: a review of the literature. Epilepsia. 1987;28 Suppl 3:S37-45. doi: 10.1111/j.1528-1157.1987.tb05776.x. PMID 3319542